CLINICAL TRIAL: NCT01934829
Title: Randomized Controlled Phase II Study of the Prophylactic Effect of Urea-Based Cream on Sorafenib-Associated Hand-Foot Skin Reactions in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Urea Cream Treatment Sorafenib-Associated HSFR in HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Anti-Cancer Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1163
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- urea-based cream (Experimental): Advanced HCC throughout China were treated with 10% urea-based cream 3 times per day plus best supportive care, starting on day 1 of sorafenib treatment, for up to 12 weeks
  Interventions: Drug: urea-based cream
- best supportive care (Placebo Comparator): BSC included the ad libitum use of non-urea-based moisturizing creams, alcohol-free moisturizer and petroleum jelly. Once HFSR occurred, patients were allowed any cream, including urea based creams, as guided by the investigator

INTERVENTIONS:
Drug: urea-based cream — urea-based cream (10% urea; Eucerin) 3 times per day plus best supportive care, starting on day 1 of sorafenib treatment, for a maximum of 12 weeks .
  BSC included the ad libitum use of non-urea-based moisturizing creams, alcohol-free moisturizer and petroleum jelly. Once HFSR occurred, patients were allowed any cream, including urea based creams, as guided by the investigator.
  Other Names: Nexavar is the brand name of sorafenib
  Arms: urea-based cream

SUMMARY:
Although sorafenib is effective and safe in patients with advanced hepatocellular carcinoma (HCC), it increases dermatologic toxicities, including hand-foot skin reaction (HFSR), which may have a negative impact on patient quality of life (QoL). Urea-based creams may have a prophylactic effect on sorafenib-induced HFSR in HCC patients.

DETAILED DESCRIPTION:
Mild hyperkeratosis is an early sign of HFSR and may sometimes be the only manifestation of sorafenib-associated HFSR. Urea is useful for the treatment of hyperkeratotic conditions and has been recommended for the treatment of multitargeted kinase inhibitor-related HFSR . To our knowledge, no randomized, controlled trials to date have evaluated treatments to prevent/palliate sorafenib-associated HFSR. We therefore tested the prophylactic effects of a urea-based cream on the incidence of HFSR associated with sorafenib treatment of patients with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

* The patients with hepatocellular carcinoma will receive sorafenib per instructions of the package insert
* The patients with hepatocellular carcinoma must be willing to participate in this study and provide the investigators with written consents;
* The patients must be willing and able to complete the biweekly visits for the first 3 months;
* The patients must be willing and able to fill in the patient's efficacy questionnaires. If the patients cannot use pens or pencils, the patient's acquaintances or the clinical staffs will complete these questionnaires based on the answers provided by the patients
* The patients must discontinue all prior cancer treatment in at least 3 weeks before enrollment;
* The patient's life expectancy is ≥3 months
* The patients must provide written informed consents

Exclusion Criteria:

* The patients participated in other clinical trials
* The patients received sorafenib therapy prior to enrollment
* The patients combined other treatment or used other biological therapy, chemotherapy, experimental treatment or radiotherapy
* The patient's sorafenib dosage exceeds 400mg, twice daily

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 871 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The incidence of all-grade HFSR | Starting sorafenib treatment within 12 weeks
Prophylactic topical application of ointment to reduce the hand-foot skin reactions in patients with hepatocellular carcinoma treated with sorafenib | Starting sorafenib treatment within 12 weeks

SECONDARY OUTCOMES:
The percentage of patients requiring sorafenib dose-reduction | Starting sorafenib treatment within 12 weeks
The percentage of patients requiring discontinuation of sorafenib therapy | starting sorafenib treatment within 12 weeks
The percentage of patients discontinuing treatment | starting sorafenib treatment within 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Long Ye, PHD, Principal Investigator — Zhongshan Hospital, Fudan University, Shanghai, China
Locations (11):
- China (11):
  - 301 Military Hospital, Beijing, China, Beijing, Beijing Municipality
  - 302 Military Hospital, Beijing, China, Beijing, Beijing Municipality
  - Union Hospital of Fujian Medical University, Fujian, China, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangdong, China, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangdong, China, Guangzhou, Guangdong
  - Heilongjiang Provincial Cancer Hospital, Heilongjiang, China, Haerbin, Heilongjiang
  - The 81 Hospital of the Chinese People's Liberation Army, Nanjing, China, Nanjing, Jiangsu
  - Jilin Provincial Tumor Hospital, Jilin, China, Changchun, Jilin
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai, Shanghai Municipality
  - Eastern Hepatobiliary Surgery Hospital of the Second Military Medical University, Shanghai, China, Shanghai, Shanghai Municipality
  - Tianjin Cancer Hospital, Tianjin, China, Tianjin, Tianjin Municipality

REFERENCES:
- [Result] Bosch FX, Ribes J, Cleries R, Diaz M. Epidemiology of hepatocellular carcinoma. Clin Liver Dis. 2005 May;9(2):191-211, v. doi: 10.1016/j.cld.2004.12.009. PMID 15831268
- [Result] Parkin DM, Bray F, Ferlay J, Pisani P. Estimating the world cancer burden: Globocan 2000. Int J Cancer. 2001 Oct 15;94(2):153-6. doi: 10.1002/ijc.1440. No abstract available. PMID 11668491
- [Result] Llovet JM, Burroughs A, Bruix J. Hepatocellular carcinoma. Lancet. 2003 Dec 6;362(9399):1907-17. doi: 10.1016/S0140-6736(03)14964-1. PMID 14667750
- [Result] Chang MH, Chen CJ, Lai MS, Hsu HM, Wu TC, Kong MS, Liang DC, Shau WY, Chen DS. Universal hepatitis B vaccination in Taiwan and the incidence of hepatocellular carcinoma in children. Taiwan Childhood Hepatoma Study Group. N Engl J Med. 1997 Jun 26;336(26):1855-9. doi: 10.1056/NEJM199706263362602. PMID 9197213
- [Result] Young JL Jr, Ries LG, Silverberg E, Horm JW, Miller RW. Cancer incidence, survival, and mortality for children younger than age 15 years. Cancer. 1986 Jul 15;58(2 Suppl):598-602. doi: 10.1002/1097-0142(19860715)58:2+3.0.co;2-c. PMID 3719551